CLINICAL TRIAL: NCT06579313
Title: Current Situation of Health Care in Women With HBV or HCV Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IN-US-987-7219
Record Dates: First submitted 2024-08-22; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: HBV; HCV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HBV cohort: 2000 HBsAg positive patients during 2016.7-2019.12
- HCV cohort: 500 HCV Ab positive and HCV RNA positive patients during 2020.7-2023.12

SUMMARY:
A multicenter, retrospective study conducted in male and female population infected with HBV or HCV in east China. HCV part, study will enroll 500 HCV antibody positive and HCV RNA positive patients during 2020.7-2023.12 and then observe the characteristics, duration from diagnosis to treatment, treatment rate and sustained virologic response (SVR12) among eligible female and male patients. HBV part, study will enroll 2000 HBsAg positive patients during 2016.7-2019.12 and then observe the clinical characteristics, natural history, duration from diagnosis to treatment, treatment rate and adherence among eligible female and male patients.

DETAILED DESCRIPTION:
Some of the sociocultural factors may prevent women infected with HBV or HCV benefiting from quality health care. Limited articles have ever reported the situation of health care in women with viral hepatitis. A previous study found that low HCV knowledge was observed in females, which was related to a lower willingness to be treated for HCV. Besides that, in other disease areas like hypertension, studies found that females have less awareness of their disease but have higher control over it compared with males. These findings might reflect the differences in health literacy levels which might influence disease outcomes, healthcare-seeking and adherence to treatment. This research aims to fill the data gaps of the gender differences in cascade of care in HBV and HCV, to facilitate patient activation, especially for women.

So far, data on the current health care status in HBV-infected women is scarce. With the expansion of treatment indications recommended by China CHB guidelines, more female patients will have the opportunity to gain timely and necessary treatment. This study will analyze the cascade of care by observing the duration from diagnosis to treatment and treatment adherence for women. And this knowledge will serve as a guide for interventions for the management of viral hepatitis, as well as effectively finding and activating patients who meet treatment criteria but are not being treated.

ELIGIBILITY:
Inclusion Criteria:

HBV Cohort -

* ≥18 years old
* serum HBsAg positive for >6 months
* Treatment naïve or,
* Patients who had been previously treated for HBV but discontinued for at least 1 year before enrollment

HCV Cohort -

* ≥18 years old
* HCV-Ab positive
* HCV RNA positive
* Treatment naïve or,
* Patients who had been previously treated for HCV with a regimen containing interferon and not had a sustained virologic response.

Exclusion Criteria:

* HBV/HCV Co-infection
* HIV
* History of hepatic decompensation or hepatocellular carcinoma
* Other carcinoma
* Other severe liver disease
* Severe Comorbidity like cardiovascular disease, diabetes etc.
* Patients who had discontinued previous HCV treatment because of an adverse event.
* Patients who had previously received any nucleotide analogue HCV NS5B inhibitor or any NS5A inhibitor
* Patients who had discontinued previous HBV treatment because of an adverse event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 HCV Ab+ and HCV RNA + patients during 2020.7-2023.12 and 2000 HBsAg+ patients during 2016.7-2019.12
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Rate in male in HBV cohort | from July 2020 to December 2023
  The treatment rate in male populations who meet treatment criteria recommended by China CHB guideline
Treatment Rate in female in HBV cohort | from July 2020 to December 2023
  The treatment rate in female populations who meet treatment criteria recommended by China CHB guideline
Treatment Rate in male in HCV cohort | from July 2016 to December 2019
  The treatment rate in male populations who meet treatment criteria recommended by China CHC guideline
Treatment Rate in female in HCV cohort | from July 2016 to December 2019
  The treatment rate in female populations who meet treatment criteria recommended by China CHC guideline

SECONDARY OUTCOMES:
Distribution of Income levels among male in HBV cohort | from July 2020 to December 2023
  categorize into 3 levels - low income (less than 50,000 CNY/year), medium income (50,000-300,000 CNY/year), high income (more than 300,000 CNY/year), in male populations infected with HBV
Distribution of Income levels among female in HBV cohort | from July 2020 to December 2023
  categorize into 3 levels - low income (less than 50,000 CNY/year), medium income (50,000-300,000 CNY/year), high income (more than 300,000 CNY/year), in female populations infected with HBV
Distribution of medical insurance type in male in HCV cohort | from July 2016 to December 2019
  categorize into 4 types - employee medical insurance, resident medical insurance, new rural cooperative medical scheme, self-pay, in male populations infected with HCV
Distribution of medical insurance type in female in HCV cohort | from July 2016 to December 2019
  categorize into 4 types - employee medical insurance, resident medical insurance, new rural cooperative medical scheme, self-pay, in male populations infected with HCV

CONTACTS AND LOCATIONS:
Overall Officials: Qing Xie, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No